CLINICAL TRIAL: NCT06616311
Title: A Prospective Study of the Efficacy of Radiofrequency Micro Needling for the Treatment of Melasma in Skin of Color.
Brief Title: Efficacy of Radiofrequency Micro Needling for the Treatment of Melasma in Skin of Color.
Acronym: SylfirmX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Benev Company, Inc. (Industry)
Responsible Party: Principal Investigator, Shilpi Khetarpal, Principal Investigator, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-649
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-12

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Intervention Model Description: Radiofrequency microneedling (RFMN) as a treatment for melasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Experimental): The target population is skin of color patients with melasma. Patients will receive 5 consecutive RFMN treatments over a period of 5 months.
  Interventions: Device: Radiofrequency microneedling

INTERVENTIONS:
Device: Radiofrequency microneedling — The target population is skin of color patients with melasma. Patients will receive 5 consecutive RFMN treatments over a period of 5 months.

SUMMARY:
The objective of this study is to test the effectiveness of radiofrequency microneedling (RFMN) as a treatment for melasma. The Investigator hypothesize that RFMN will be an effective treatment for melasma in skin of color patients.

DETAILED DESCRIPTION:
The target population is skin of color patients with melasma. Patients will receive 3 consecutive RFMN treatments over a period of three months. Baseline melasma severity will be measured by the modified Melasma Area and Severity Index (mMASI) score. Endpoints will be mMASI scores at 1 and 3 months post-procedure. Patient reported outcomes will be measured using the melasma quality of life (MelasQOL) validated patient questionnaire at screening and at both follow up visits. The long-term goal of future studies would be to provide melasma patients, particularly those with skin of color, with improved therapeutic options for the treatment of their melasma, as compared to current treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, at least 18 years of age
* Fitzpatrick skin types IV-VI
* Clinically diagnosed melasma
* No topicals (retinol, vitamin C serum, etc) for 6 weeks before Visit 1 (with exception of sunscreen)

Exclusion Criteria:

* is currently pregnant or planning to conceive during the study period
* is using topical or oral therapy or other treatment for melasma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy as determined by change in mMASI scoring of melasma severity post-treatment. | 9 months
  The primary endpoint is treatment efficacy as determined by change in mMASI scoring of melasma severity post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

DOCUMENTS (1):
  • Study Protocol (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT06616311/Prot_001.pdf